CLINICAL TRIAL: NCT05708456
Title: Investigation of the Effect of the Mobile Application Developed for the Management of Symptoms in Hypothyroid Patients
Brief Title: The Effect of Mobile Application on Hypothyroid Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SakaryaU,
Record Dates: First submitted 2022-12-22; First posted 2023-02-01 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-12

CONDITIONS: Hypothyroidism; Symptom Management; Symptoms and Signs; Mobile Application; Digital Health
MeSH Terms: conditions — Hypothyroidism; Signs and Symptoms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Application of data collection forms for the initial evaluation. Teaching the use of the mobile application, monitoring the use of the mobile application in the experimental group by the researcher for 12 weeks, and applying the data collection forms to the patients in the 6th and 12th weeks.
  Interventions: Other: Mobile application with symptom management
- Control Group (No Intervention): Application of data collection forms for the initial evaluation. Application of data collection forms to the patients in the 6th and 12th weeks. No intervention will be made to the patients in the control group other than the routine service provided in the outpatient clinic.

INTERVENTIONS:
Other: Mobile application with symptom management — In this study, patients will be given evidence-based advice via a mobile application to manage their symptoms.
  Arms: Intervention Group

SUMMARY:
Hypothyroidism refers to the common pathological condition of thyroid hormone deficiency. The annual incidence of hypothyroidism is 3.5 per 1000 in women and 0.6 in per 1000 men. Hypothyroidism is seen 5-8 times more frequently in women than in men. Patients with hypothyroidism have a higher prevalence of cardiovascular risk factors and often have metabolic syndrome features such as hypertension, increased waist circumference, and dyslipidemia. Other signs and symptoms include bradycardia, slow speech, swelling in the eyes and face, weight gain, decreased sweating, hair loss, pallor, forgetfulness, decreased concentration, depression, irritability, tongue growth, loss of appetite, palpitations, decreased hearing, menstrual irregularities, muscle pains, and cramps. Depending on all these signs and symptoms, hypothyroidism can negatively affect the quality of life of individuals. Therefore, it is essential to reduce symptoms and to improve patients' abilities to manage them. It is stated that the appropriate use of mobile health applications helps the patient to make informed decisions about health management and treatment. Therefore, this study plans to investigate the effect of mobile technology on symptom management in individuals with hypothyroidism, whose symptoms range from mild to severe.

DETAILED DESCRIPTION:
The research will be carried out in Sakarya University Training and Research Hospital Endocrinology Polyclinic. It is planned to include a total of 80 patients in the research (40 patients in the control group - 40 patients in the experiment group). The first step of this study is to develop the scales to be used in the study. The Hypothyroidism Symptom Management Scale and the Hypothyroidism Symptom Severity Scale will be developed. In the second stage, data will be collected. The Patient Information Form, Hypothyroidism Symptom Severity Scale, and Hypothyroidism Symptom Management Scale will be applied to the experimental group that meets the research criteria and agrees to participate. The patient's blood test findings (TSH, T3, T4, Anti-Tg, Anti TPO, Antithyroglobulin, Hmg, Hct) will also be recorded at the first meeting. The researcher will measure the patient's height, weight, and vital signs. The mobile application will be introduced to the patients and downloaded to the patient's phones, and a username and password will be created. The content of this mobile application; Interventions will be planned based on evidence-based practices to alleviate or reduce the symptoms of hypothyroidism. These initiatives are planned both in written form and in short video narration. Patients will be asked to watch the videos in the mobile application for the first week. At the end of each week, patients will be asked to report symptoms in the application and read and follow the recommendations for the relevant symptom. The usage period of the mobile application is determined as three months (12 weeks). In addition, at the end of the fourth week, patients will be followed up by having the symptom management scale and symptom severity scale applied via the mobile application. In the 6th and 12th weeks, evaluations of the patient's laboratory test results, vital signs, height, and weight measurements, will also be evaluated besides the scales. In the first interview with the individuals in the control group, after explanations are made about the research and their verbal and written consents are accordingly obtained, First, the Patient Information Form, the Hypothyroidism Symptom Severity Scale, and the Hypothyroidism Symptom Management Scale will be administered as a pre-test. At the first interview, the patient's blood test findings, height, weight, and vital signs will be recorded. Measurements will be repeated when individuals come to their outpatient clinic appointments 6 and 12 weeks after the first interview.

ELIGIBILITY:
Inclusion Criteria:

* Able to communicate,
* Who agrees to participate in the study,
* Able to use a mobile phone with android or ıos (iPhone os) operating system
* No vision and dexterity problems,
* Without communication difficulties and cognitive impairment,
* Literate
* Being diagnosed with hypothyroidism

Exclusion Criteria:

* Pregnant patients,
* Those with a diagnosed psychiatric illness,
* Those who use antidepressants,
* Patients who experienced trauma or an acute illness during the study (12 weeks)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-02-15 (Estimated); Primary Completion 2023-09-17 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Symptom management scale | Change from day 1 to week 12 of the study.
  To detect an increase in scores on the HypothyroidismSymptom management scale at Week 12 compared to baseline.
Symptom Severity scale | Change from day 1 to week 12 of the study
  To detect a decrease in the score on the Symptom Severity scale at week 12 compared to baseline.

SECONDARY OUTCOMES:
Thyroid function (Only TSH) | Change from day 1 to week 12 of the study.
  The effect of the patient's thyroid function tests on the 12th week compared to the baseline.
  Blood test (Only TSH) will be performed during the outpatient follow-up at the first, sixth, and 12th weeks.
Blood lipid (LDL) | Change from day 1 to week 12 of the study
  The effect on the patient's blood lipid profile [LDL cholesterol (low-density lipoprotein)] levels compared to baseline at week 12. Blood tests will be performed during the outpatient follow-up at the first, sixth, and 12th weeks.
Blood lipid (HDL) | Change from day 1 to week 12 of the study
  The effect on the patient's blood lipid profile [HDL cholesterol (high-density lipoprotein)] levels compared to baseline at week 12. Blood tests will be performed during the outpatient follow-up at the first, sixth, and 12th weeks.
Blood lipid (total cholesterol ) | Change from day 1 to week 12 of the study
  The effect on the patient's blood lipid profile (Total cholesterol) levels compared to baseline at week 12. Blood tests will be performed during the outpatient follow-up at the first, sixth, and 12th weeks.
Blood pressure | Change from day 1 to week 12 of the study
  The effect on the patient's blood pressure values compared to the baseline at the 12th week.The researcher will measure it.
Body Mass Index | Change from day 1 to week 12 of the study
  The effect on the patient's Body Mass Index compared to baseline at week 12. The researcher will measure it. Body Mass Index is calculated by dividing the person's weight in kilograms by the square of the person's height in meters (kg/m²).

CONTACTS AND LOCATIONS:
Locations (1):
- Seyma Trabzon, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No